CLINICAL TRIAL: NCT00994500
Title: A Phase I Study of Vorinostat and Bortezomib in Children With Refractory or Recurrent Solid Tumors, Including CNS Tumors and Lymphomas
Brief Title: Vorinostat and Bortezomib in Treating Young Patients With Refractory or Recurrent Solid Tumors, Including Central Nervous System Tumors and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01980; ADVL0916; CDR0000656719; COG-ADVL0916; U01CA097452 (NIH)
Record Dates: First submitted 2009-10-10; First posted 2009-10-14 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Childhood Burkitt Lymphoma; Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Germ Cell Tumor; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Medulloepithelioma; Childhood Meningioma; Childhood Mixed Glioma; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Childhood Oligodendroglioma; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Central Nervous System Embryonal Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Malignant Germ Cell Tumor; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Burkitt Lymphoma; Choroid Plexus Neoplasms; Lymphoma, Large B-Cell, Diffuse; Meningioma; Lymphoma, Extranodal NK-T-Cell; Oligodendroglioma; Lymphoma, Large-Cell, Anaplastic; Astrocytoma; Familial ependymoma; Dendritic Cell Sarcoma, Interdigitating; Medulloblastoma; Optic Nerve Glioma; Recurrence | interventions — Vorinostat; Bortezomib

ARMS (1):
- Treatment (vorinostat, bortezomib) (Experimental): Patients receive oral vorinostat once daily on days 1-5 and 8-12 and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat; Drug: bortezomib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with bortezomib in treating young patients with refractory or recurrent solid tumors, including CNS tumors and lymphoma. Vorinostat and bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose and/or recommended phase II dose of vorinostat in combination with bortezomib in pediatric patients with refractory or recurrent solid tumors, including central nervous system tumors and lymphoma.

II. To define and describe the toxicities of this regimen in these patients. III. To characterize the pharmacokinetics of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of this regimen within the confines of a phase I study.

II. To assess the biologic activity of bortezomib by measuring NF-κB activity in peripheral blood mononuclear cells (PBMC).

III. To assess the biologic activity of bortezomib by measuring endoplasmic reticulum stress response using the GRP78 molecular chaperone marker in PBMC.

OUTLINE: This is a multicenter, dose-escalation study of vorinostat.

Patients receive oral vorinostat once daily on days 1-5 and 8-12 and bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and during course 1 of study for further analysis.

After completion of study therapy, patients are followed up within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors, including CNS tumors or lymphoma

  * Histological confirmation not required for the following diagnoses

    * Intrinsic brain stem tumors
    * Optic pathway gliomas
    * Pineal tumors and elevations of cerebral spinal fluid or serum tumor markers, including alpha-fetoprotein or beta-human chorionic gonadotropin, allowed
    * Relapsed or refractory disease
* Must have measurable or evaluable tumor
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky performance status (PS) 60-100% for patients > 16 years of age OR Lansky PS60-100% for patients ≤ 16 years of age

  * Neurologic deficits inpatients with CNS tumors must have been relatively stable for a minimum of 1week
  * Patients who are unable to walk because ofparalysis, but who are up in a wheelchair, will be considered ambulatory for thepurpose of assessing the performance score
* ANC ≥ 1,000/μL
* Platelet count ≥ 100,000/μL (transfusion independent, defined as not receiving platelet transfusions within the past 7 days)

  * Patients with known bone marrow metastatic disease allowed provided they meet the blood count criteria and are not known to be refractory to platelet transfusion
* Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)

  * Patients with known bone marrow metastatic disease allowed provided they meet the blood count criteria and are not know to be refractory to RBC or platelet transfusion
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age and/or gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 (male) or 1.4 (female) (13 to < 16 years of age)
  * 1.7 (male) or 1.4 (female) ( ≥ 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 times upper limit ofnormal
* ALT ≤ 110 U/L
* Serum albumin ≥ 2 g/dL
* QTc interval ≤ 450 milliseconds
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to swallow capsules or liquids
* Able to comply withthe safety-monitoring requirements of the study, in the opinion of the investigator
* No peripheral neuropathy ≥ grade 2 within the past 14 days
* No known hypersensitivity to vorinostat or bortezomib
* No uncontrolled infection
* No concurrent enzyme-inducing anticonvulsants
* Must be recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* More than 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)
* At least 7 days since prior therapy with any of the following:

  * Hematopoietic growth factors
  * Biologic (anti-neoplastic) agent

    * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Corticosteroids unless on a stable or decreasing dose
* At least 7 days or 3 half-lives, whichever is longer, since prior monoclonal antibodies
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior total-body irradiation therapy, craniospinal radiotherapy, or ≥ 50% of pelvis irradiated
* At least 6 weeks since prior substantial bone marrow radiotherapy
* At least 3 months since prior stem cell transplantation or rescue and no evidence of active graft-vs-host disease
* At least 2 weeks since prior and no concurrent valproic acid
* At least 6 weeks since priorimmunotherapy (e.g., tumor vaccines)
* No prior vorinostat
* No other concurrent investigational drugs or other anticancer agents, including chemotherapy, radiotherapy, immunotherapy, or biologic therapy

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose defined as the maximum dose at which fewer than one-third of patients experience DLT according to NCI CTCAE version 3.0 | 21 days
  In addition to determination of the MTD, a descriptive summary of all toxicities will be reported.

SECONDARY OUTCOMES:
Disease response assessed according to RECIST criteria | Up to 30 days
  Will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Muscal, Principal Investigator — COG Phase I Consortium
Locations (6):
- United States (6):
  - Childrens Memorial Hospital, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas